CLINICAL TRIAL: NCT02511626
Title: Quality of Life in Endometriosis - a Case Control Study Using Internationally Validated Questionnaires
Brief Title: Quality of Life in Endometriosis - a Case Control Study
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Triemli Hospital (Other); Cantonal Hospital of St. Gallen (Other); Kantonsspital Baden (Other); Kantonsspital Winterthur KSW (Other); Kantonsspital Schaffhausen (Unknown); Charite University, Berlin, Germany (Other); University Hospital, Aachen (Other); Vivantes Kliniken Berlin (Unknown); Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Endo_QOL
Record Dates: First submitted 2015-07-20; First posted 2015-07-30 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Endometriosis; Quality of Life; Pain; Sexuality; Anxiety; Depression; Infertility
Keywords: endometriosis; quality of life; professional activity; pain; infertility; sexuality; partnership; anxiety; depression; stress; childhood trauma; medical support; dyspareunia
MeSH Terms: conditions — Endometriosis; Pain; Sexuality; Anxiety Disorders; Depression; Infertility; Dyspareunia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Case group: Women with a surgically confirmed diagnosis of endometriosis
- Control group 1: Women without any evidence of endometriosis (= no clinical symptom and/or no surgical evidence of endometriosis)
- Control group 2: Women without endometriosis (surgically confirmed) but chronic abdominal/pelvic pain due to other reasons (e.g. Crohn's disease, colitis etc)

SUMMARY:
Endometriosis, one of the most common diseases of women during their reproductive period., may present a chronic disabling disease with major impact on women's life. Therapeutic options are limited and recurrence of disease symptoms is frequent.

The current study investigates the quality of life and several risk factors for the development of endometriosis as well as satisfaction with medical support in a minimum of 600 women with different stages of endometriosis and the same number of control women matched for age (± 3 years) and nationality. To evaluate specific features of endometriosis-associated pain a second group of 100 women with chronic abdominal/pelvic pain not related to endometriosis is investigated. Recruitment takes place in different university clinics, and districts hospitals in Switzerland, Germany. And Austria. Control women i.e. women without any evidence for endometriosis presenting for annual routine gynaecological controls are collected at the same places.

A composition of different internationally validated questionnaires as well as specific questions on dealing with endometriosis is used to collect information on the quality of life and potential risk factors for endometriosis. Questions on sexuality and partnership are also distributed to women's partners. All diagnosis of endometriosis and classification of ASRM (American Society for Reproductive Medicine) disease stages are based on woman's medical charts.

DETAILED DESCRIPTION:
With a prevalence of 7-10% endometriosis is one of the most common diseases of women during their reproductive period. There is a broad range of clinical symptoms of endometriosis, which may vary between an incidental asymptomatic finding and a chronic severely painful disease. Symptoms are nearly independent from disease stage and current therapeutic options do not permit to reliably reduce symptoms to an acceptable level. Independent from the therapy chosen, about 20% of women re-develop clinical symptoms in the first year and another 50% within a period of five years.

The currently provided medical support concentrates on surgical and medical i.e. hormonal options. Although it seems evident that endometriosis-associated pain will have a serious impact on the daily life of women attaint and there is a broad literature on the effect of other chronic pain diseases on patients' lives, comparable data for endometriosis are rare. Also, support models to allow women to integrate a chronic endometriosis into their daily life are currently lacking. To provide a reliable basis for the development of better holistic support models, the current study collects data on different aspects of the quality of life in a minimum of 600 women with different stages of endometriosis and a minimum of 600 control women matched for age (± 3 years) and nationality. To evaluate which features of the quality of life are specific for endometriosis a second control group of 100 women with chronic abdominal/pelvic pain not related to endometriosis is investigated. Recruitment takes place in different university clinics, and districts hospitals in Switzerland, Germany and Austria. Control women i.e. women without any evidence for endometriosis presenting for annual routine gynaecological controls are collected at the same places.

A composition of different internationally validated questionnaires as well as specific questions on dealing with endometriosis is used to collect information on the quality of life and potential risk factors for endometriosis. The questionnaire includes basic socio-demographic data, life style parameters, a general as well as gynaeco-obstetric history including detailed questions on the diagnosis, treatment and current symptoms of endometriosis. In addition questionnaires on pain (modified version of the Brief Pain Inventory (BPI), Pain Disability Index (PDI), resources (SOC), stress perception (PSQ20), professional development, satisfaction with medical support, adverse childhood experiences (modified version of the childhood trauma questionnaire (CTQ), daily life, partnership (Partnerschaftsfragebogen, PFB), sexuality (modified version of the Brief Index of Sexual Functioning and Global sexual functioning) and anxiety/depression (PHQ, GAD) have to be completed by study participants. Socio-demographic questions, questions on partnership as well as on the estimated impact of endometriosis on partnership /sexuality were also given to study participants' partners. In addition to the current quality of life potential risk factors for the development of endometriosis e.g. traumatic childhood experiences are evaluated as well as satisfaction with medical support are evaluated.

All diagnosis of endometriosis and classification of ASRM disease stages are based on woman's medical charts.

ELIGIBILITY:
Inclusion Criteria:

female >18 years fluent German

* Cases: diagnosis of endometriosis Control 1: no endometriosis, no chronic pain Control 2: no endometriosis, chronic abdominal/pelvic pain

Exclusion Criteria:

* male (Except for partner questionnaires)
* <18years
* not fluent in German

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female Age >18
  Case group: women with endometriosis Healthy volunteers in control group
Sampling Method: Probability Sample
Enrollment: 1267 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Quality of life i.e. pain, infertility, partnership, sexuality, depression, anxiety, stress, medical support, comorbidities and risk factors in the development of endometriosis: childhood trauma, life style factors, menstrual history | The questionnaire is answered once after at inclusion in the study, different questions cover different time periods ranging from childhood (0-17 years) to the actual situation (last 4 weeks/ 24hours) as specified in the questionnaire
  The outcome measures are assessed with internationally validated questionnaires i.e. modified version of the Brief Pain Inventory and Pain Disability Index, modified Form des Childhood Trauma Questionnaire, Brief Symptom Inventory, partnership questionnaire (PFB), modified version of the Brief Index of Sexual Functioning und Global sexual functioning, Hospital Anxiety and Depression Scale (HADS) as well as the questionnaire on life satisfaction (FLZ)

SECONDARY OUTCOMES:
Prevalences of diseases such as dyspareunia, sexual disorders or adverse childhood experiences in the control group. | Once at inclusion in the study
  Measurements with internationally validated questionnaires and womens' medical history according to medical charts
Comorbidity of chronic pain. | Once at inclusion in the study
  Measurements with internationally validated questionnaires and womens' medical history according to medical charts

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Leeners, Prof. Dr., Principal Investigator — Clinic for Reproductive Endocrinology, University Hospital Zurich, Switzerland
Locations (1):
- Clinic for Reproductive Endocrinology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Candan A, Kohl Schwartz A, Birchler K, Leeners B. Psychosomatic comorbidity in endometriosis: A multi-center, cross-sectional study identifying an underestimated factor in current medical support. J Psychosom Res. 2025 Sep;196:112346. doi: 10.1016/j.jpsychores.2025.112346. Epub 2025 Aug 9. PMID 40815907
- [Derived] El Hadad S, Schwartz ASK, Gassner C, Haeberlin F, von Orelli S, Imesch P, Leeners B. Partnership and relationship happiness in endometriosis related chronic pelvic pain: a multicenter case-control study. Front Psychol. 2024 Oct 14;15:1382067. doi: 10.3389/fpsyg.2024.1382067. eCollection 2024. PMID 39469237
- [Derived] El-Hadad S, Lasser D, Sachs MK, Schwartz ASK, Haeberlin F, von Orelli S, Eberhard M, Leeners B. Dysmenorrhea in adolescents requires careful investigation of endometriosis-an analysis of early menstrual experiences in a large case-control study. Front Reprod Health. 2023 Aug 25;5:1121515. doi: 10.3389/frph.2023.1121515. eCollection 2023. PMID 37693279
- [Derived] Sperschneider ML, Hengartner MP, Kohl-Schwartz A, Geraedts K, Rauchfuss M, Woelfler MM, Haeberlin F, von Orelli S, Eberhard M, Maurer F, Imthurn B, Imesch P, Leeners B. Does endometriosis affect professional life? A matched case-control study in Switzerland, Germany and Austria. BMJ Open. 2019 Jan 9;9(1):e019570. doi: 10.1136/bmjopen-2017-019570. PMID 30782670
- [Derived] Ramin-Wright A, Schwartz ASK, Geraedts K, Rauchfuss M, Wolfler MM, Haeberlin F, von Orelli S, Eberhard M, Imthurn B, Imesch P, Fink D, Leeners B. Fatigue - a symptom in endometriosis. Hum Reprod. 2018 Aug 1;33(8):1459-1465. doi: 10.1093/humrep/dey115. PMID 29947766
- [Derived] Liebermann C, Kohl Schwartz AS, Charpidou T, Geraedts K, Rauchfuss M, Wolfler M, von Orelli S, Haberlin F, Eberhard M, Imesch P, Imthurn B, Leeners B. Maltreatment during childhood: a risk factor for the development of endometriosis? Hum Reprod. 2018 Aug 1;33(8):1449-1458. doi: 10.1093/humrep/dey111. PMID 29947745
- [Derived] Kohl Schwartz AS, Wolfler MM, Mitter V, Rauchfuss M, Haeberlin F, Eberhard M, von Orelli S, Imthurn B, Imesch P, Fink D, Leeners B. Endometriosis, especially mild disease: a risk factor for miscarriages. Fertil Steril. 2017 Nov;108(5):806-814.e2. doi: 10.1016/j.fertnstert.2017.08.025. PMID 29079275